CLINICAL TRIAL: NCT01322984
Title: Cognitive and Emotional Processing of Social Stimuli in Children and Youth With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Tromso (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010/238
Record Dates: First submitted 2011-03-02; First posted 2011-03-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Startle
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal controls (Active Comparator): Normal children and youths
  Interventions: Behavioral: Pictures; Behavioral: Startle eliciting noise
- ASD (Experimental): Children and youths diagnosed with autism spectrum disorder (ASD)
  Interventions: Behavioral: Pictures; Behavioral: Startle eliciting noise

INTERVENTIONS:
Behavioral: Pictures — The participants will be exposed to pictures of faces and non-facial stimuli presented on a PC screen.
Behavioral: Startle eliciting noise — Startle will be elicited by 95 dB noise, presented at different times after picture onset.

SUMMARY:
Children and youth diagnosed with autism spectrum disorder (ASD) have been shown to react abnormally to social stimuli, especially to human faces. Children and youth with ASD show less interest in social stimuli, and may even avoid looking at or interact with such stimuli. It has been proposed that social stimuli elicit reactions like fear and stress in individuals with ASD, and this explains the lack of interest and avoidance. The present project investigates this hypothesis.

ELIGIBILITY:
For ASD group:

Inclusion Criteria:

* Diagnosed with autism spectrum disorders

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The eyeblink of the Startle reflex is measured. | The startle reflex will be measured in relation to picture presentations during the experiment (e.g. day 1).
  The startle reflex is potentiated when participants are influenced by negative emotions. Accordingly, startle will be measured in relation to picture presentation to gauge the emotional effect of the pictures. It is expected that the ASD group will show fear potentiated startle to pictures of human faces.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, University of Tromso, Tromsø, Troms, Norway

REFERENCES:
- See also: Related Info — http://uit.no